CLINICAL TRIAL: NCT00385411
Title: Therapeutic Follow-up Observational Study and Population Kinetics Ancillary Study of Valproate Microgranules (Micropakine® SR) in Patients Aged Between 6 Months and 15 Years Suffering From Epilepsy.
Brief Title: Study of Valproate in Young Patients Suffering From Epilepsy
Acronym: VAPOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: "Medical Affairs Study Director", sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8971; EudraCT #: 2005-004041-33
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- valproate (Experimental)
  Interventions: Drug: valproate microgranules

INTERVENTIONS:
Drug: valproate microgranules — 20 to 30 mg/kg/day

SUMMARY:
Main objective: Therapeutic follow-up study Evaluate the clinical and biological safety of valproate administered as microgranules, under standard prescription conditions, with therapeutic follow-up and individual dosage adjustment, using valproate plasma concentrations and antiepileptic comedication as well as biological assays.

Secondary objectives: Ancillary population kinetics study

* Estimate the pharmacokinetic parameters of valproate administered as microgranules under standard therapeutic conditions within the population studied, from the therapeutic follow-up data.
* Evaluate the influence of individual characteristics on the pharmacokinetic parameters.
* Describe the relationship between plasma concentrations and adverse events for valproate and the main anti-epileptic comedications.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 months and 15 years.
* Suffering from any type of epilepsy.
* Receiving at the time of inclusion valproate in the form Micropakine® SR 20 to 30 mg/kg/d by oral route, in 2 daily administrations and at most two other antiepileptic drugs (an antiepileptic benzodiazepine treatment taken daily or on demand more than 2 times weekly, must be considered as an antiepileptic treatment).
* Followed by hospital paediatricians or neuropaediatricians.
* For whom the consent has been signed by the parents or the holders of parental authority and if possible by the child him/herself.
* For whom the parents or legal guardian do not have any language or cultural obstacle for understanding the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2006-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Clinical and biological safety. | at each visit
Pharmacokinetic parameters and covariables likely to explain the variability in the pharmacokinetic parameters of valproate | Ancillary population kinetics study

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France